CLINICAL TRIAL: NCT00150319
Title: An Open-Label Study To Assess The Pharmacokinetics, Safety And Toleration Of Vfend®; Iv Containing Sbecd As An Excipient Following Multiple Dosing With Vfend®; I.V. In Subjects With Moderately Impaired Renal Function
Brief Title: An Open-Label Study To Assess The Pharmacokinetics, Safety And Toleration Of Vfend®; Following Multiple Dosing With Vfend
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: See Detailed Description
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: A1501070
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2008-09-29 (Estimated); Status verified 2008-09

CONDITIONS: Kidney Failure
MeSH Terms: conditions — Renal Insufficiency | interventions — Voriconazole

INTERVENTIONS:
Drug: Vfend®; I.V.

SUMMARY:
This is a study to investigate the pharmacokinetics, safety and tolerability of intravenous voriconazole and SBECD in patients with moderate renal insufficiency

DETAILED DESCRIPTION:
The study was put on hold after the first subject was enrolled and experienced a serious adverse event (SAE) of renal failure chronic after receiving his I.V. dose on Day 1. The study was taken off hold after the subject recovered and an independent consultant had deemed the SAE as not treatment related; however, the site was unwilling to enroll additional subjects. Another site, based in New Orleans, was damaged by hurricane Katrina and was unable to enroll any subjects. A decision was made by the sponsor to terminate the study on 11 Apr 2006 due to poor study enrollment. There were no safety or efficacy concerns regarding the study in the decision to terminate the trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate renal insufficiency

Exclusion Criteria:

* Active infection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2005-06; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Ability to tolerate up to seven days of intravenous voriconazole without worsening of pre-existing renal insufficiency

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United States (4):
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, Minneapolis, Minnesota
  - Pfizer Investigational Site, Knoxville, Tennessee
  - Pfizer Investigational Site, Austin, Texas

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1501070&StudyName=An+Open%2DLabel+Study+To+Assess+The+Pharmacokinetics%2C+Safety+And+Toleration+Of+Vfend%26%23174%3B+Following+Multiple+Dosing+With+Vfend